CLINICAL TRIAL: NCT06131632
Title: Conserving Surgery in Inflammatory Breast Cancer After Neoadjuvant Chemotherapy in Patients With Clinical Complete Response (ConSIBreC): a Randomized Clinical Trial
Brief Title: Conserving Surgery in Inflammatory Breast Cancer After Neoadjuvant Chemotherapy
Acronym: ConSIBreC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Consibrec Trial
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Breast Cancer
Keywords: inflammatory breast cancer; breast conserving surgery; radical mastectomy
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — Mastectomy, Segmental; Mastectomy, Modified Radical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast conserving surgery (Experimental)
  Interventions: Procedure: Breast conserving surgery
- Radical modified mastectomy (Active Comparator)
  Interventions: Procedure: Radical modified mastectomy

INTERVENTIONS:
Procedure: Breast conserving surgery — Remove only a small part of the breast
  Arms: Breast conserving surgery
Procedure: Radical modified mastectomy — Remove all the breast parenchyma, nipple and skin
  Arms: Radical modified mastectomy

SUMMARY:
Inflammatory breast cancer is an aggressive and rare form of breast cancer, which accounts for 2-3% of all breast cancers. The classic presentation of inflammatory breast cancer includes erythema, edema, and peau d'orange of at least one/third of the breast.

Current treatment of inflammatory breast cancer include: neoadjuvant chemiotherapy, modified radical mastectomy and radiation therapy.

In the last two decades the development of new targeted therapies has significantly improved the efficacy of neoadjuvant chemiotherapy allowing a de-escalation of surgical treatment in patients with non-inflammatory breast cancer that achieve clinical complete response.

There are few retrospective studies that evaluate implications of surgical treatment on survival among these patients. This may justify trial aims to investigate the possible use of the breast conserving surgery in patients with inflammatory breast cancer that achieve clinical complete response after neoadjuvant chemiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory breast cancer
* Clinical complete response after neoadjuvant chemiotherapy
* Targeted tumor
* Written informed consent

Exclusion Criteria:

* Metastasis
* Progression disease
* Recurrent disease
* Contraindications to adjuvant radiation therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
local recurrence rate | 24 months
  Rate of recurrence in the breast parenchyma after conserving surgery vs radical mastectomy

SECONDARY OUTCOMES:
local recurrence-free survival | 24 months
  Rate of disease free survival after breast conserving surgery vs radical mastectomy
overall survival | 24 months
  overall survival after breast conserving surgery vs radical mastectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS,, Roma, Italy